CLINICAL TRIAL: NCT04050397
Title: Exercise Intervention to Reduce Adverse Quality of Life Effects From Androgen Deprivation Therapy for Prostate Cancer - Randomized Clinical Trial
Brief Title: Exercise and Quality of Life During Androgen Deprivation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Varalan urheiluopisto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Patient School 1
Record Dates: First submitted 2018-06-27; First posted 2019-08-08 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
Keywords: androgen deprivation therapy; exercise; quality of life; blood glucose; cholesterol; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participant will be randomized 1:1 to either supervised exercise for 12 weeks or to follow given exercise program on their own.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised exercise arm (Experimental): Informational initiation lecture and supervised exercise twice a week for 12 weeks followed by 12 weeks of non-supervised exercise.
  Interventions: Other: Progressive supervised weight training; Other: Lecture
- Non-supervised exercise arm (Active Comparator): Informational initiation lecture and only non-supervised exercise
  Interventions: Other: Lecture

INTERVENTIONS:
Other: Progressive supervised weight training — 12 weeks of progressive weight training twice a week supervised by a qualified physiotherapist.
  Arms: Supervised exercise arm
Other: Lecture — Urologist informs participants on adverse effects of castration treatments and benefits of regular exercise. Physiotherapist gives an exercise program to follow at home, and nutritionist informs patients on correct nutrition to assist physical exercise.

SUMMARY:
This study evaluates effects of supervised exercise in reducing adverse effects of hormonal treatment, increasing quality of life and in inducing a long-term change into more active lifestyle in prostate cancer patients on androgen deprivation therapy. All participants will attend a starting lecture at the beginning of the trial, after which they are randomly allocated to attend 3 months of either supervised or non-supervised exercise program. Leisure time activity, quality of life, blood sugar and cholesterol values, and body composition of participants will be evaluated at three time-points; at recruitment, after 12 weeks and after 24 weeks. Effects on quality of life will also be qualitatively evaluated with single- and group interviews.

DETAILED DESCRIPTION:
Androgen deprivation therapy (ADT) is commonly used in management of advanced or recurrent prostate cancer. It also frequently used adjuvant to curative-intent radiation therapy for localized prostate cancer. Low testosterone levels during androgen deprivation commonly cause adverse effects reducing quality of life. Most common adverse effects include fatigue, weight gain, loss of lean muscle mass, hyperglycemia and hypercholesterolemia.

Regular exercise, especially programs involving combination of both aerobic exercise and resistance training has been shown to reduce to reduce adverse effects of ADT on physical functioning and quality of life. It may also improve disease prognosis.

The study compares effects of supervised and unsupervised exercise on plasma lipid parameters (total cholesterol, LDL, HDL and triglycerides) and glucose levels (fasting plasma glucose, glycated hemoglobin), overall quality of life and on average daily exercise activity in men with prostate cancer and under ADT. As secondary outcome we will study effect on continued exercise activity after the intervention, changes in body composition, blood pressure and risk of fractures, castration resistance as well as death due to prostate cancer and due to any cause.

Study hypothesis is that supervised exercise will improve quality of life, lipid and glucose parameters and increase daily exercise activity more that non-supervised exercise. We also expect higher continued exercise activity, greater changes in body composition and blood pressure and lowered risk of fractures and death in the supervised exercise group.

This is a randomized, controlled clinical trial. The study aims to recruit 40 men on ADT for prostate cancer. This will be a pilot study to estimate effect sizes in Finnish population to inform further larger trial.

All participants attend introductory lecture, where a urologist informs them about adverse effects of ADT and positive effects of exercise during ADT, exercise instructor gives advice for training both at home and in the gym and nutritional therapeutist tells about nutrition to overcome adverse effects of ADT and support training.

After the introductory lecture the participants are randomized 1:1 to either the supervised or non-supervised exercise group (Figure). Men in the supervised group participate in progressive group exercise sessions twice a week for total of 12 weeks at the Varala sports academy in Tampere, Finland. Each exercise session includes both aerobic and resistance training targeting all major muscle groups (Additional document I, exercise program). The non-supervised group will exercise independently for 12 weeks according to the instructions given at the introductory lecture. The first control visit will be after this first period of 12 weeks of exercise.

After the first follow-up visit both group will continue non-supervised exercise for 12 weeks, after which the second control visit will be arranged. Special focus on the second control visit is to see how many in each group has been able to carry on active exercising, i.e. has the intervention promoted long-term change in exercise activity.

Both study group will be given Polar wrist activity monitors to be used 24 h/day for the entire course of the study.

All participants are asked to fill validated quality of life surveys EORTC QLQC-30 (overall quality of life) and EORTC QLQC-PR25 (prostate cancer-specific quality of life) at baseline and again at 1st and 2nd control visits. Additionally, qualitative evaluation of quality of life as well as perceived possibilities and obstacles for exercise are evaluated in individual- and group interviews during the study visits. Plasma lipid and glucose parameters, blood pressure and body composition will be measured at each of these visits.

At each visit a separate blood sample is taken and stored for future measurement of biomarkers associated with prostate cancer progression, glucose and lipid metabolism and effects of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing castration treatment for prostate cancer
* Informed consent for the study

Exclusion Criteria:

* Unable to participate in exercise (ECOG 2 or greater)
* High bone fracture risk (as judged by the primary physician)
* Unable to understand spoken and written instructions in Finnish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-08-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Daily total activity | At randomization and twice more at 12 week intervals
  Daily activity as measured by wrist activity monitor worn by the participants at all times during the study. Measured as metabolic equivalents of task (MET) units. Range from 0.9 to 23.
Fasting plasma total cholesterol | At randomization and twice more at 12 week intervals
  Value measure in mmol/l
Fasting plasma LDL cholesterol | At randomization and twice more at 12 week intervals
  Value measure in mmol/l
Fasting plasma HDL cholesterol | At randomization and twice more at 12 week intervals
  Value measure in mmol/l
Fasting plasma triglycerides | At randomization and twice more at 12 week intervals
  Value measure in mmol/l
Fasting plasma glucose level | At randomization and twice more at 12 week intervals
  Value measured in mmol/l
Blood glycated hemoglobin (HbA1C) level | At randomization and twice more at 12 week intervals
  Value measured in mmol/mol
Overall quality of life | At randomization and twice more at 12 week intervals
  Score from validated survey EORTC QLQ-C30, score range from 0-100, with 100 denoting the highest quality of life
Prostate cancer-specific quality of life | At randomization and twice more at 12 week intervals
  Score from validated survey EORTC QLQ-PR25, score range from 0-100, with 100 denoting the highest quality of life

SECONDARY OUTCOMES:
Change in daily activity after the intervention | Measured daily for 12 weeks' time after the intervention
  Change in daily activity of the supervised exercise group after completion of 12 weeks of supervised exercise as measured by wrist activity monitor in MET units, range from 0.9 to 23.
Subjective adverse effects of castration treatment | At randomization and twice more at 12 week intervals
  The effect of supervised exercise on subjective adverse effects of castration treatment for prostate cancer. Qualitative assessment in three individual interviews and one group interview. No scaling used as this is a qualitative rather than quantitative end-point
Lean body mass | At randomization and twice more at 12 week intervals
  Bioimpedance-based measurement of lean body mass as percentage of total body mass measured with TANITA MC-780 device
Muscle mass | At randomization and twice more at 12 week intervals
  Bioimpedance-based measurement of muscle mass as percentage of total body mass measured with TANITA MC-780 device
Skeletal mass | At randomization and twice more at 12 week intervals
  Bioimpedance-based measurement of skeletal mass as percentage of total body mass measured with TANITA MC-780 device measured with TANITA MC-780 device
Fat mass | At randomization and twice more at 12 week intervals
  Bioimpedance-based measurement of fat mass as percentage of total body mass measured with TANITA MC-780 device measured with TANITA MC-780 device
Metabolic age | At randomization and twice more at 12 week intervals
  Metabolic age measured with bioimpedance-based TANITA MC-780 device
Systolic blood pressure | At randomization and twice more at 12 week intervals
  Value measured in mmHg
Diastolic blood pressure | At randomization and twice more at 12 week intervals
  Value measured in mmHg

OTHER OUTCOMES:
Time to castration resistance | Followed yearly for up to 15 years from randomization
  Time to castration resistance as defined by two consecutive rising PSA levels and increase of 50% or more from the nadir. Measured as months between the study recruitment and first record of castration resistance. Information obtained from patient files.
Time to death | Followed yearly for up to 15 years from randomization
  Time to death due to any cause. Measured as months between the study recruitment and date of death. Information obtained from patient files and national death certificate registry.
Time to prostate cancer death | Followed yearly for up to 15 years from randomization
  Time to death due to prostate cancer. Measured as months between the study recruitment and date of death. Information obtained from patient files and national death certificate registry.
Bone fractures | Followed yearly for up to 15 years from randomization
  Occurrence of any bone fracture requiring either conservative or operative management. Information obtained from patient files and national hospital discharge registry. Fracture site and it's management are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Teemu Murtola, MD PhD, Principal Investigator — Tampereen University, Faculty of Medicine and Health Technology
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared since it is prohibited by the ethics board and by patient consent

REFERENCES:
- [Derived] Rantaniemi L, Jussila I, Siltari A, Ahtiainen JP, Hakulinen A, Harju E, Sormunen J, Nordstrom T, Tammela TLJ, Murtola TJ. Is Exercise During Androgen Deprivation Therapy Effective and Safe? A Randomized Controlled Trial. Scand J Med Sci Sports. 2025 Jun;35(6):e70084. doi: 10.1111/sms.70084. PMID 40481694

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT04050397/Prot_SAP_000.pdf